CLINICAL TRIAL: NCT00399685
Title: Study to Evaluate the Effect of Efavirenz Coadministration on the Pharmacokinetics of the Active Moieties of a Combined Oral Contraceptive Containing Ethinyl Estradiol and Norgestimate in Healthy Female Subjects
Brief Title: Drug Interaction - Oral Contraceptive
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: AI266-145
Record Dates: First submitted 2006-11-14; First posted 2006-11-15 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: HIV Infections
Keywords: HIV
MeSH Terms: conditions — HIV Infections | interventions — Moxifloxacin; efavirenz

ARMS (4):
- A (Active Comparator)
  Interventions: Drug: Ortho Tri-Cyclen LO
- B (Active Comparator)
  Interventions: Drug: Ortho Cyclen
- C (Active Comparator)
  Interventions: Drug: Ortho Cyclen + Efavirenz
- D (Active Comparator)
  Interventions: Drug: Ortho Cyclen

INTERVENTIONS:
Drug: Ortho Tri-Cyclen LO — Tablets, oral, OTC Lo 1 tab/daily (no dosage units), once daily, 28 days.
  Arms: A
Drug: Ortho Cyclen — Tablet, oral, Ortho Cyclen 1 tab/daily (no dosage units), once daily, 28 days.
  Arms: B
Drug: Ortho Cyclen + Efavirenz — Tablet, oral, OC + EFV 600 mg, once daily, 14 days.
  Other Names: Sustiva
  Arms: C
Drug: Ortho Cyclen — Tablet, oral, OC 1 tab daily (no dosage units), once daily, 7 days.
  Arms: D

SUMMARY:
The purpose of this study is to administer a combined oral contraceptive containing ethinyl estradiol and norgestimate with the HIV treatment of efavirenz to healthy females in order to assess if the concentrations of the oral contraceptives change. The safety of this treatment regimen will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Women of childbearing potential with intact ovarian function who have been on a stable method of oral contraceptives for at least 2 months prior to the start of the study.
* Documented acceptable Pap smear within 1 year of the start of the study
* BMI of 18-32 kg/m²

Exclusion Criteria:

* Males
* Subjects with abnormal menstrual cycle within 2 months prior to the start of the study
* History of conditions in which oral contraceptives are contraindicated
* History of migraine with focal aura
* History of uncontrolled hypertension
* Positive screening test for HIV-1,-2, HIV viral RNA, Hepatitis B surface antigen, or Hepatitis C antibody
* History of diagnosed mental illness or suicidal ideation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2006-12; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
To determine the effect coadministration of efavirenz 600 mg on the pharmacokinetics of ethinyl estradiol and the metabolite of norgestimate | throughout the study

SECONDARY OUTCOMES:
Characterize the pharmacokinetics of efavirenz coadministered with the oral contraceptive Ortho Cyclen | throughout the study
Assess the effect of efavirenz coadministered with Ortho Cyclen on serum progesterone levels | throughout the study
Assess the safety of efavirenz coadministered with Ortho Cyclen | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Covance Clinical Research Unit San Diego, San Diego, California
  - Northwest Kinetics, Tacoma, Washington